CLINICAL TRIAL: NCT03172065
Title: The Effect of Adding Intrathecal Dexmedetomidine on Shoulder Tip Pain During Laparoscopic Ovarian Cystectomy Under Bupivacaine Spinal Anaesthesia. Randomised Controlled Study.
Brief Title: Dexmedetomidine and Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, Lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDGL
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia Complication
MeSH Terms: interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): will receive 3.5 ml (17.5 mg) hyperbaric Bupivacaine + 0.5 ml saline
  Interventions: Drug: Normal saline
- Dexmedetomidine group (Other): will receive 3.5 ml (17.5 mg) hyperbaric Bupivacaine + 0.5 ml dexmedetomidine (0.5 mic)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Normal saline — intravenous flluid
  Arms: control group
Drug: Dexmedetomidine — anaesthetic adjuvants and pain killer medication.
  Arms: Dexmedetomidine group

SUMMARY:
Conventionally General anaesthesia remains the choice for the majority of open abdominal surgical procedures, and regional anaesthesia is preferred only for patients who are at high risk under general anaesthesia . The main reason for selecting spinal anaesthesia as the first choice for laparoscopic cases was its advantages over general anaesthesia which include uniform total muscle relaxation, a conscious patient, economical, relatively uneventful recovery, pain free early postoperative period and the protection from potential complications of general anaesthesia. The main debatable point, however, seems to be the status of respiratory parameters among the two modes of anaesthesia during laparoscopic surgery. In this context it can be stated that spontaneous physiological respiration during spinal anaesthesia would always be better than an assisted respiration as in general anaesthesia.

The pneumo-peritoneum induced rise in intra-abdominal pressure including pressure on the diaphragm and carbon dioxide induced peritoneal irritation are the factors to be considered

ELIGIBILITY:
Inclusion Criteria:

* Elective gynaecological laparoscopic surgery
* Age 20-45 yrs
* Suspected surgery time 30 minutes
* Inflation pressure <13 Cm H20

Exclusion Criteria:

* Contraindications to regional block (infection at the needle insertion site)
* Altered conscious level.
* Pregnancy
* Body mass index >35
* Height <155 cm
* Patients who have difficulty understanding the study protocol

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
occurrence shoulder tip pain | 48 hours

SECONDARY OUTCOMES:
intraoperative haemodynamic stability, et co2, sao2. | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided